CLINICAL TRIAL: NCT03208036
Title: Restoration of Cognitive Function With TDCS and Training in Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D0180-R; I01RX000180 (NIH)
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Results first posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-11

CONDITIONS: Schizophrenia; Bipolar Disorder; Schizo Affective Disorder
Keywords: schizophrenia; tdcs; working memory; cognitive remediation; cognition; serious mental illness
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Psychotic Disorders | interventions — Transcranial Direct Current Stimulation; Cognitive Remediation

STUDY DESIGN:
Intervention Model Description: This is a double-blind, double-baseline, sham-controlled study in which participants are randomized to receive either tDCS or sham stimulation concurrent with cognitive training.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, interventionists, and the outcome assessors will be blind to participant condition. The neuromodulation device can be pre-programmed to deliver either tDCS or sham stimulation when an ID code is entered. The study personnel randomizing participants and programming the equipment will not have contact with participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TDCS (Experimental): TDCS offered concurrent with working memory focused cognitive training
  Interventions: Device: TDCS; Behavioral: Cognitive Remediation; Behavioral: Bridging Group
- Sham (Sham Comparator): Sham stimulation offered concurrent with working memory focused cognitive training
  Interventions: Device: Sham Stimulation; Behavioral: Cognitive Remediation; Behavioral: Bridging Group

INTERVENTIONS:
Device: TDCS — 1 mA of anodal stimulation will be applied to the left dorsal lateral cortex (F3) concurrent with working memory focused cognitive training for 20 minutes
  Other Names: Transcranial Direct Current Stimulation
  Arms: TDCS
Device: Sham Stimulation — Participants will receive 20 seconds of 1 mA anodal stimulation applied to the left dorsal lateral cortex (F3) concurrent with working memory focused cognitive training to mimic the effect of the active condition
  Other Names: Sham
  Arms: Sham
Behavioral: Cognitive Remediation — Participants complete 60 minutes of computer-based cognitive training. All tasks are adaptable in terms of difficulty and require working memory skills. Sessions always begin with N-back and complex span tasks completed concurrent with tDCS or sham stimulation. Other tasks selected from Happy Neuron software and experimental working memory tasks are used throughout the protocol.
Behavioral: Bridging Group — Participants complete 45 minutes of activities and discussion to practice engaging cognitive skills through performance of everyday activities and to learn strategies to use cognitive abilities most effectively. Curriculum generated from Action-based Cognitive Remediation and Compensatory Cognitive Training intervention manuals.

SUMMARY:
Development of interventions that can effectively target and remediate the cognitive and functional impairment associated with serious mental illness is a treatment priority. Transcranial direct current stimulation (tDCS) is a safe, non-invasive neuromodulation technique that is capable of stimulating brain activity to facilitate learning. The primary objective of this study is to evaluate the pairing of two therapeutic techniques, cognitive remediation and tDCS, as a cognitively enhancing intervention. This study is designed to test the hypotheses that cognitive remediation paired with tDCS will be more efficacious than cognitive remediation delivered with sham stimulation and that intervention-induced cognitive change will be sustainable.

To examine the incremental benefit of pairing tDCS with cognitive remediation, clinically stable outpatients between the ages of 18-65 who have a diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder will be enrolled in a double-blind, double-baseline, sham-controlled clinical trial. Participants will be randomized in a 1:1 ratio to receive either tDCS or sham stimulation concurrent with working memory focused cognitive remediation. Training will be offered to participants in a small group format. Training will consist of 48 sessions, with 2-3 sessions scheduled in a week. Each training session will last 2 hours. One hour will be spent completing cognitive exercises that require working memory skills on a computer. TDCS or sham stimulation will be offered concurrent with the first 20 minutes of training with a StarStim neuromodulator. One mA of anodal stimulation will be applied to the left dorsal lateral prefrontal cortex and the cathodal electrode will be placed in the contralateral supraorbital position. Upon completion of working memory training, participants will transition to a 45-minute bridging group focus on application of cognitive skills in everyday life. To assess intervention-induced change, working memory, other aspects of cognition, functional capacity, community functioning, and symptom severity will be assessed pre- and post-intervention. Sustainability of intervention-induced change will be assessed with an assessment session 6 weeks post-intervention. Mixed effect, repeated measure ANOVAS will be used to analyze intervention-induced change.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible for the study if they have a diagnosis of schizophrenia, schizoaffective disorder, or bipolar I disorder and are clinically stable at the time of enrollment

  * defined as not severely depressed or acutely manic and no hospitalizations or antipsychotic medication changes in the four weeks prior to enrollment

Exclusion Criteria:

* Met criteria for a severe alcohol or substance use disorder in the last 6 months
* Met criteria for a mild alcohol or substance use disorder in the last month
* A history of head injury or neurological disease that has compromised cognitive functioning
* Ability to speak English is not sufficient to understand study procedures
* Diagnosis of learning disability, mental retardation, or pervasive developmental disorder
* Diagnosis of a medical condition that is incompatible with tDCS procedures
* Participant does not demonstrate understanding of study procedures during the consent process
* A documented history of behavioral problems that prevent participation in a group intervention
* Participated in a study of tDCS or cognitive remediation in the previous 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tasha M Nienow, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared. Final data set will be made available upon written request. In order to fulfill requests, I will ensure that all data storage locations are kept current in the Minneapolis VAHCS Data Inventory database, and I will store all study research records and data for a minimum of 6 fiscal years post study closure.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available at study closure and accessible for 6 years.
Access Criteria: When a request for data is received, an agreement will be set up and approved by the local facility before data is released.

RESULTS

PARTICIPANT FLOW:
Period: Baseline Assessment
Arm/Group | TDCS | Sham
Started | 11 | 11
Completed | 10 | 10
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: 2nd Baseline Assessment
Arm/Group | TDCS | Sham
Started | 10 | 10
Completed | 9 | 8
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Intervention
Arm/Group | TDCS | Sham
Started | 9 | 8
Completed | 6 | 6
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2
Period: 4-month Assessment
Arm/Group | TDCS | Sham
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: 5.5 Month Assessment
Arm/Group | TDCS | Sham
Started | 6 | 6
Completed | 5 | 4
Not Completed | 1 | 2
Not completed — Partial data collected due to COVID-19 pandemic and remote procedures only | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TDCS | Sham | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.55 (8.29) | 51.27 (7.94) | 51.41 (8.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 8 | 11 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 8 | 7 | 15
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 22
Years of Education [Mean (Standard Deviation); unit: years] | 13.27 (1.42) | 13.46 (1.04) | 13.37 (1.23)
Test of Premorbid Functioning Standard Score [Mean (Standard Deviation); unit: units on a scale] — This is a measure of intellectual function prior to the onset of illness or disease. Scores range from 50 to 135. Higher scores indicate better intellectual functioning. A score of 100 is considered average.
  units on a scale | 94.09 (12.23) | 96.79 (8.30) | 95.44 (10.27)
N-Back D-Prime Score [Mean (Standard Deviation); unit: D prime] — This is a working memory task. A 2-back version was administered. D prime a measure of response accuracy that takes into account both hit rate and false alarm rate was used to measure performance. Scores range from -4.54 to 4.54, with higher, positive scores indicating better working memory performance. A score of 0 indicates chance level performance. Population: 5 participants withdrew from the baseline assessment process before data on this measure could be collected from them.
  D prime
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 1.07 (.74) | 1.15 (.47) | 1.11 (.61)

OUTCOME MEASURES:

1. Primary Outcome: Working Memory Capacity Composite Score
Description: This is a measure of one core component of working memory. Proportion correct average from Change Detection and Change Localization Tasks. Score ranges from 0.00 to 1.00, with a higher score indicating better performance
Time Frame: Total score at Baseline, 4 months, and 5.5 months
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: Proportion of correct responses
Arm/Group | TDCS | Sham
Number analyzed (Participants) | 6 | 6
Proportion of correct responses
  Baseline | .64 (.13) | .70 (.07)
  4-month assessment | .64 (.13) | .72 (.05)
  5.5 month assessment | .63 (.08) | .71 (.05)
Statistical Analysis 1: Comparison: TDCS vs Sham; Mixed effect, repeated measure ANOVA to assess change between baseline, 4-month, and 5.5 month assessments. Test for a Group x Time interaction; Test type: Superiority; p = .69, Mixed Models Analysis
Statistical Analysis 2: Comparison: TDCS vs Sham; Mixed effect, repeated measure ANOVA to assess change between baseline, 4-month, and 5.5 month assessments. Test for a Main Effect of Time; Test type: Superiority; p = .74, Mixed Models Analysis

2. Primary Outcome: Goal Maintenance Composite Score
Description: This is a measure of one core component of working memory. Performance on the Dot Pattern Expectancy Task and AX-Continuous Performance Task was measured with d prime. D Prime is a measure of response accuracy that takes into account both hit rate and false alarm rate. This measure of response accuracy ranges from -4.546 to 4.546, with a higher score indicating better performance. A score of 0 indicates chance level performance. D prime scores reflecting overall performance on the Dot Pattern Expectancy Task and the AX-Continuous Performance Task were averaged. The resulting d prime score reflects performance on the goal maintenance component of working memory.
Time Frame: D Prime at Baseline, 4 months, and 5.5 months
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: D Prime
Arm/Group | TDCS | Sham
Number analyzed (Participants) | 6 | 6
D Prime
  Baseline | 3.34 (.58) | 2.91 (1.94)
  4-months | 2.78 (1.36) | 2.71 (1.50)
  5.5 months | 2.60 (.48) | 2.73 (1.38)
Statistical Analysis 1: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .62, Mixed Models Analysis
Statistical Analysis 2: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .24, Mixed Models Analysis

3. Primary Outcome: Interference Control Composite Score
Description: This is a measure of one core component of working memory. Performance on Rotation and Reading Complex Span Tasks was measured with z-scores. Scores range from -3 to 3, with a higher positive score indicating better performance. A score of 0 represents the sample mean at the baseline assessment. The z-scores reflecting overall performance on Rotation and Reading Span Tasks were averaged to create one z-score that reflects performance on the interference control component of working memory.
Time Frame: Z-score at Baseline, 4 months, and 5.5 months
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | TDCS | Sham
Number analyzed (Participants) | 6 | 6
Z-score
  Baseline | -.37 (.62) | -.20 (.94)
  4-month assessment | -.03 (.52) | -.10 (1.16)
  5.5-month assessment | -.28 (.80) | -.40 (.94)
Statistical Analysis 1: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .47, Mixed Models Analysis
Statistical Analysis 2: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .09, Mixed Models Analysis
Statistical Analysis 3: Comparison: TDCS; Within group change assessed between baseline and 4-month assessment; Test type: Superiority; p = .02, t-test, 2 sided
Statistical Analysis 4: Comparison: TDCS; Within group change assessed between baseline and the 5.5 month assessment; Test type: Superiority; p = .48, t-test, 2 sided
Statistical Analysis 5: Comparison: Sham; Within group change assessed between baseline and 4-month assessment; Test type: Superiority; p = .66, t-test, 2 sided
Statistical Analysis 6: Comparison: Sham; Within group change assessed between baseline and 5.5 month assessment; Test type: Superiority; p = .46, t-test, 2 sided

4. Primary Outcome: The University of California San Diego Performance-Based Skills Assessment Total Score
Description: This is a performance-based measure of functional capacity to perform activities of daily living. This measure has two scales, measuring financial and communication skills. The two scales are summed to create a total score. The Total score ranges from 0-100, with a higher score indicating better performance.
Time Frame: Total score at Baseline, 4 months, and 5.5 months
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TDCS | Sham
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 78.33 (9.73) | 73.67 (14.95)
  4-month assessment | 82.00 (9.55) | 76.50 (11.42)
  5.5 month assessment | 78.36 (13.67) | 77.76 (9.34)
Statistical Analysis 1: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .68, Mixed Models Analysis
Statistical Analysis 2: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .45, Mixed Models Analysis

5. Secondary Outcome: First-Episode Social Functioning Scale Actual Performance Total Score
Description: Total score summed from Actual Performance subscales 1-5. This is a self-report measure of social and community functioning in the past 3 months. Scores reflect the frequency with which participants report engaging in a behavior. Total score ranges from 20-80, with a higher score indicating better social functioning in the community.
Time Frame: Total score at Baseline, 4 months, and 5.5 months
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TDCS | Sham
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 55.33 (5.43) | 55.17 (8.68)
  4-month assessment | 56.17 (5.42) | 56.50 (8.53)
  5.5 month assessment | 58.67 (10.17) | 53.50 (8.17)
Statistical Analysis 1: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .81, Mixed Models Analysis
Statistical Analysis 2: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .31, Mixed Models Analysis

6. Secondary Outcome: Novel N-Back Task D Prime Score
Description: This is a working memory task. The number and picture n-back tasks are novel versions of the training tasks used in this protocol. D-prime, a measure of response accuracy that takes into account hit rate and false alarm rate was used to measure overall performance on each task. This measure of performance accuracy ranges from -4.546 to 4.546, with a higher, positive score indicating better performance. A score of 0 indicates chance level performance. D prime scores from the number and picture task were average to create one d prime measure that reflects performance on novel, untrained n-back measures. Improvement on these tasks would indicate generalization of learning from the trained tasks.
Time Frame: D prime at Baseline, 4 months, and 5.5 months
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: D prime
Arm/Group | TDCS | Sham
Number analyzed (Participants) | 6 | 6
D prime
  Baseline | 1.24 (.46) | 1.29 (.46)
  4-month assessment | 1.41 (.62) | 1.34 (.46)
  5.5 month assessment | 1.42 (.30) | 1.33 (.19)
Statistical Analysis 1: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .79, Mixed Models Analysis
Statistical Analysis 2: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .50, Mixed Models Analysis

7. Secondary Outcome: Complex Span Task Z-score
Description: This is a working memory task. This measure is an indicator of whether participants were able to improve on a task procedurally similar to the training tasks. Rotation and Reading complex span tasks are novel versions of training tasks. A z-score was used to measure performance on each task. Z-scores range from -3 to 3, with a higher positive score indicating better performance. A score of 0 represents the sample mean at the baseline assessment. Z-scores from the Rotation and Reading span tasks were averaged to create one measure of working memory. Improvement on this task would indicate generalization of learning from the training.
Time Frame: Z-score at Baseline, 4 months, and 5.5 months
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | TDCS | Sham
Number analyzed (Participants) | 6 | 6
Z-score
  Baseline | -.37 (.62) | -.20 (.94)
  4-month assessment | -.03 (.52) | -.10 (1.16)
  5.5 month assessment | -.28 (.80) | -.40 (.94)
Statistical Analysis 1: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .47, Mixed Models Analysis
Statistical Analysis 2: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .09, Mixed Models Analysis
Statistical Analysis 3: Comparison: TDCS; Within group change assessed between baseline and 4-month assessment; Test type: Superiority; p = .02, t-test, 2 sided
Statistical Analysis 4: Comparison: TDCS; Within group change assessed between baseline and the 5.5 month assessment; Test type: Superiority; p = .48, t-test, 2 sided
Statistical Analysis 5: Comparison: Sham; Within group change assessed between baseline and 4-month assessment; Test type: Superiority; p = .66, t-test, 2 sided
Statistical Analysis 6: Comparison: Sham; Within group change assessed between baseline and the 5.5 month assessment; Test type: Superiority; p = .46, t-test, 2 sided

8. Secondary Outcome: MATRICS Consensus Cognitive Battery Processing Speed Subscale and the Reasoning and Problem-Solving Subscale T-score Average
Description: Two subscales from the MATRICS Consensus Cognitive Battery, the Processing Speed subscale and the Reasoning and Problem-Solving subscale, were averaged to create a composite that reflects performance on cognitive functions closely related to working memory. Performance on each subscale was measured with a T-score. T-scores range from 0-100. A score of 50 reflects the population mean, with a standard deviation of 10. On each subscale, a higher score indicated better performance in the cognitive domain. Improvement on this composite T-score would indicate generalization of training gains to untrained cognitive domains.
Time Frame: T-score at Baseline, 4 months, and 5.5 months
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | TDCS | Sham
Number analyzed (Participants) | 6 | 6
T-score
  Baseline | 44.58 (10.17) | 49.92 (10.47)
  4-month assessment | 43.50 (8.39) | 49.17 (9.42)
  5.5 month assessment | 44.15 (10.35) | 50.04 (7.92)
Statistical Analysis 1: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .99, Mixed Models Analysis
Statistical Analysis 2: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .84, Mixed Models Analysis

9. Secondary Outcome: Brief Psychiatric Rating Scale Total Score
Description: This is a 24-item measure of psychiatric symptom severity. Each item is rated on a 1-7 scale, with a higher score indicating that the symptom is more severe. Brief Psychiatric Rating Scale Total score can range from 24-168, with a higher score indicating the presence of more severe psychiatric symptoms.
Time Frame: Total score at Baseline, 4 months, and 5.5 months
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TDCS | Sham
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 34.00 (3.03) | 43.50 (16.53)
  4-month assessment | 32.00 (3.69) | 38.00 (9.12)
  5.5 month assessment | 31.83 (3.37) | 43.17 (11.89)
Statistical Analysis 1: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .25, Mixed Models Analysis
Statistical Analysis 2: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .08, Mixed Models Analysis
Statistical Analysis 3: Comparison: TDCS; Within group change assessed between baseline and 4-month assessment; Test type: Superiority; p = .14, t-test, 2 sided
Statistical Analysis 4: Comparison: TDCS; Within group change assessed between baseline and 5.5-month assessment; Test type: Superiority; p = .02, t-test, 2 sided
Statistical Analysis 5: Comparison: Sham; Within group change assessed between baseline and 4-month assessment; Test type: Superiority; p = .24, t-test, 2 sided
Statistical Analysis 6: Comparison: Sham; Within group change assessed between baseline and 5.5-month assessment; Test type: Superiority; p = .93, t-test, 2 sided

10. Secondary Outcome: Brief Negative Symptom Severity Scale Total Score
Description: This is a 13-item scale that measures the severity of negative symptoms. Each item is rated from 0-6, with a higher score indicating that the symptom is more severe. Brief Negative Symptom Severity Scale Total score can range from 0 to 78, with a higher score indicating more severe negative symptoms
Time Frame: Total score at Baseline, 4 months, and 5.5 months
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TDCS | Sham
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 18.50 (7.97) | 25.17 (14.41)
  4-month assessment | 13.83 (6.74) | 21.17 (8.28)
  5.5 month assessment | 14.40 (7.61) | 21.00 (9.12)
Statistical Analysis 1: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .98, Mixed Models Analysis
Statistical Analysis 2: Comparison: TDCS vs Sham; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = .08, Mixed Models Analysis
Statistical Analysis 3: Comparison: TDCS; Within group change assessed between baseline and 4-month assessment; Test type: Superiority; p = .08, t-test, 2 sided
Statistical Analysis 4: Comparison: TDCS; Within group change assessed between baseline and 5.5-month assessment; Test type: Superiority; p = .06, t-test, 2 sided
Statistical Analysis 5: Comparison: Sham; Within group change assessed between baseline and 4-month assessment; Test type: Superiority; p = .28, t-test, 2 sided
Statistical Analysis 6: Comparison: Sham; Within group change assessed between baseline and 5.5-month assessment; Test type: Superiority; p = .23, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events between July 2018 and December 2021. Individual participants were enrolled in the study and monitored for adverse events for as long as 10 months.
Arm/Group | TDCS | Sham
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TDCS (N=9) | Sham (N=8)
Hospitalization (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Participant was hospitalized for treatment and stabilization of a pre-existing medical condition while enrolled in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT03208036/Prot_SAP_000.pdf